CLINICAL TRIAL: NCT05771727
Title: Impact of Covid-19 Pandemic on Children With Neuromuscular Disease and Their Parents in Turkey: Parent Perspective
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Bora, Physiotherapist, Hacettepe University
Other Study IDs: GO 21/722
Record Dates: First submitted 2023-03-14; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of children with pediatric neuromuscular diseases: Parents of a total of 169 children with pediatric neuromuscular diseases, including 63 Duchnenne Muscular Dystrophy, 53 Spinal Muscular Atrophy and 18 other pediatric neuromuscular diseases (Congenital Muscular Dystrophy, Hereditary Motor and Sensory Neuropathy, Becker Muscular Dystrophy, Limb-Girdle Muscular Dystrophy, etc.) were included in the study
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — The 55-item survey created by the researchers was applied online to determine the psychological and physical effects of COVID-19 on neuromuscular patients and their families. This survey also included the Content of the 9-Item Caregiver COVID-19 Limitations Scale (CCLS-9).

SUMMARY:
Parents of children with neuromuscular disease have been already at risk of depression, anxiety and burden. Additionally, the daily lives of children with neuromuscular disease and their parents have been significantly affected by the COVID-19 pandemic. Therefore, this study investigated parents' perspective on the effect of the COVID-19 pandemic on children with neuromuscular diseases and themselves.

DETAILED DESCRIPTION:
The 55-item survey created by the researchers was applied online to determine the psychological and physical effects of COVID-19 on neuromuscular patients and their families. This survey also included the Content of the 9-Item Caregiver COVID-19 Limitations Scale (CCLS-9).

ELIGIBILITY:
Inclusion Criteria:

* taking care for a child with NMD whose age was between 0-18 years,
* having the ability to read and write Turkish language,
* having access to phone or e-mail,
* being volunteer.

Exclusion Criteria:

* having a child who have an additional diagnosis besides NMD and taking care of any other person in the family.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children with pediatric neuromuscular diseases
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
The questionnaire which created by the researchers | 30 minutes
  The 55-item survey created by the researchers was applied online to determine the psychological and physical effects of COVID-19 on neuromuscular patients and their families.

SECONDARY OUTCOMES:
Content of the 9-Item Caregiver COVID-19 Limitations Scale (CCLS-9) | 5 minutes
  This scale consists of 9 items and has a scoring system between 1-10 for each item which is chosen by the caregiver. According to the CCLS-9 scale, the lowest anxiety, stress or burden of the caregiver scored as 1 while the highest level was 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided